CLINICAL TRIAL: NCT02485873
Title: REal-LIfe Evidence on Stroke Prevention in Patients With Atrial Fibrillation
Brief Title: Real-Life Evidence on Stroke Prevention in SPAF
Acronym: RELIEF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: 18073; DBOX 2014/00799 (Other: Company internal)
Record Dates: First submitted 2015-05-28; First posted 2015-06-30 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Atrial Fibrillation (Prevention of Stroke)
Keywords: Non-valvular atrial fibrillation (NVAF); Pevention; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban: Non-valvular Atrial Fibrillation (NVAF) patients who were initiated on rivaroxaban for stroke prevention
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Vitamin K antagonists (VKA): NVAF patients who were initiated on VKA (predominately phenprocoumon in Germany) for stroke prevention
  Interventions: Drug: Vitamin K antagonists

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — As prescribed by treating physicians
  Groups: Rivaroxaban
Drug: Vitamin K antagonists — As prescribed by treating physicians
  Groups: Vitamin K antagonists (VKA)

SUMMARY:
To obtain a better understanding on the comparative effectiveness of rivaroxaban and vitamin K antagonists (VKA) for stroke prevention in patients with non-valvular atrial fibrillation (SPAF) in a real-life setting

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years on the day of the first prescription of the study drug (= index date) during study selection window
* Diagnosis of NVAF on start date of study or anytime during 365 days before this date
* Availability of follow-up at least 180 days after the date of the first prescription of study drug within selection window of study (exposure start date)
* Evidence of patient activity in the database during 90 days before the date of the first prescription of target drug within selection window.

Exclusion Criteria:

* Patients with valvular AF
* Prescriptions of Oral Anticoagulants (OACs): VKA, Dabigatran, Rivaroxaban before index date
* Prescription of more than one OAC on the index date or switch to another OAC during the follow-up period
* Prescriptions of < 15mg rivaroxaban at index date or during the follow-up period for patients in rivaroxaban cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation (NVAF)
Sampling Method: Non-Probability Sample
Enrollment: 8607 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of any of the following: Ischemic stroke (IS), Transient ischemic attack (TIA), Intracerebral hemorrhage (IH), Other non-traumatic intracranial hemorrhage including subdural hemorrhage, Myocardial infarction (MI) | Within 1 year after treatment start
  Composite cardiovascular endpoint

SECONDARY OUTCOMES:
Time to first occurrence of IS | Within 1 year after treatment start
  Single cardiovascular event
Time to first occurrence of TIA | Within 1 year after treatment start
  Single cardiovascular event
Time to first occurrence of IH | Within 1 year after treatment start
  Single cardiovascular event
Time to first occurrence of Other non-traumatic intracranial hemorrhage including subdural hemorrhage | Within 1 year after treatment start
  Single cardiovascular event
Time to first occurrence of MI | Within 1 year after treatment start
  Single cardiovascular event
Incidence density in study population of IS | Within 1 year after treatment start
Incidence density in study population of TIA | Within 1 year after treatment start
Incidence density in study population of IH | Within 1 year after treatment start
Incidence density in study population of Other non-traumatic intracranial hemorrhage including subdural hemorrhage | Within 1 year after treatment start
Incidence density in study population of MI | Within 1 year after treatment start
Incidence density in study population of any of the following: IS, TIA, IH, Other non-traumatic intracranial hemorrhage including subdural hemorrhage, MI | Within 1 year after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany